CLINICAL TRIAL: NCT04130438
Title: Efficacy of Medical Therapy in Women and Men With Angina and Myocardial Bridging
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment, insufficient funding
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jennifer A Tremmel, MD, MS, Interventional cardiologist, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 47447
Record Dates: First submitted 2019-04-01; First posted 2019-10-17 (Actual); Results first posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Myocardial Bridging
MeSH Terms: conditions — Myocardial Bridging | interventions — Nebivolol; Diltiazem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Beta Blocker (nebivolol) (Active Comparator)
  Interventions: Drug: Nebivolol
- Calcium Channel Blocker (diltiazem) (Active Comparator)
  Interventions: Drug: Diltiazem
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Nebivolol — The intervention to be tested is oral beta blocker (nebivolol 2.5 mg) vs. calcium channel blocker (Diltiazem-SR 120 mg) vs. placebo. Once enrolled, baseline data will be gathered and subjects will be randomly assigned to a treatment arm. Subjects will be instructed to take their assigned study drug once a day for 30 days.
  Arms: Beta Blocker (nebivolol)
Drug: Diltiazem — The intervention to be tested is oral beta blocker (nebivolol 2.5 mg) vs. calcium channel blocker (Diltiazem-SR 120 mg) vs. placebo. Once enrolled, baseline data will be gathered and subjects will be randomly assigned to a treatment arm. Subjects will be instructed to take their assigned study drug once a day for 30 days.
  Arms: Calcium Channel Blocker (diltiazem)
Other: Placebo — The intervention to be tested is oral beta blocker (nebivolol 2.5 mg) vs. calcium channel blocker (Diltiazem-SR 120 mg) vs. placebo. Once enrolled, baseline data will be gathered and subjects will be randomly assigned to a treatment arm. Subjects will be instructed to take their assigned study drug once a day for 30 days.
  Arms: Placebo

SUMMARY:
The proposed clinical trial is relevant to public health because it is expected to expand the differential diagnosis and provide an evidence--based therapy for the large population of patients with angina in the absence of obstructive CAD who currently remain undiagnosed and untreated. It, therefore, upholds an important part of the mission of the The National Heart, Lung, and Blood Institute (NHLBI), which is to promote the treatment of heart disease and enhance the health of all individuals so that they can live longer and more fulfilling lives.

DETAILED DESCRIPTION:
Angina in the absence of obstructive coronary artery disease (CAD) affects millions, resulting in a reduced quality of life and a burden on the health care system. Previous work has focused on endothelial and microvascular dysfunction as causes of angina in these patients, but even when these etiologies are tested for, nearly half of patients remain undiagnosed, and proven therapies are lacking. The long--term goal of this research proposal is to improve the lives of patients with angina in the absence of obstructive CAD. These patients have been found to have a disproportionate prevalence of myocardial bridges (MBs) (60% vs. 30% in the general population).

MBs are known to cause angina, and the mechanism by which they do so is also known, but MBs have not been actively studied in the context of patients with angina in the absence of obstructive CAD. Medical therapies for symptomatic MBs, including beta blockers and calcium channel blocker have been suggested, but have never been appropriately tested, and may not be better than placebo. The overall objective of this research proposal is to demonstrate that MBs are an important and treatable cause of angina in patients with non--obstructive CAD.

The investigator will conduct the first--ever randomized, double--blind, placebo--controlled trial of medical therapy in patients with angina and an MB. The rationale is that a proven treatment would significantly expand the paradigm by which patients with angina in the absence of obstructive CAD are evaluated and treated. Our central hypothesis is that beta blockers and calcium channel blockers are effective treatments for reducing angina in patients with an MB compared with placebo. Guided by strong preliminary data, this hypothesis will be tested by pursuing two specific aims: 1) Determine the efficacy of beta blockers and calcium channel blockers in treating patients with angina and an MB and 2) Identify predictors of efficacy of beta blockers and calcium channel blockers in treating patients with angina and an MB. For Aim #1, the investigator will randomize a total of 360 adult patients with angina and an MB into one of three treatment arms: beta blocker (nebivolol), calcium channel blocker (diltiazem), or placebo (1:1:1).

Efficacy will be determined after 30 days on the study drug by a change in angina, as assessed by the Seattle Angina Questionnaire (SAQ). The investigator will also evaluate changes in exercise capacity, as well as drug adherence and side effects. For Aim #2, the investigator will evaluate MB muscle index (MMI, a product of MB length x depth) by coronary computed tomography angiography, as well as male sex, as predictors of efficacy. Randomization will be stratified on sex, ensuring a balance of women and men in each arm. The proposed research is innovative because it shifts the current clinical perspective on angina in the absence of obstructive CAD by considering myocardial bridging as a potential etiology.

It is also significant because it will substantially increase the number of patients with angina in the absence of obstructive CAD that clinicians are able to diagnose and treat, ultimately leading to improvements in quality of life and a reduction in health care costs.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥18 years
2. Stable angina (typical or atypical, based on Diamond criteria (35))
3. Exercise stress echocardiogram or exercise stress test (with beta blocker or calcium channel blocker held) performed within six months of enrollment
4. CCTA or invasive coronary angiogram confirming the presence of an MB
5. Absence of obstructive CAD, as demonstrated by no ischemia on stress testing and no significant obstructive CAD (coronary stenosis <50%) on CCTA or invasive coronary angiogram

Exclusion Criteria:

1. Asymptomatic
2. Status--post heart transplant
3. Presence of another likely explanation of chest pain, such as pulmonary hypertension, hypertrophic obstructive cardiomyopathy, or aortic stenosis
4. Presence of an acute coronary syndrome (unstable angina, NSTEMI, or STEMI), Tako--tsubo, or cardiogenic shock
5. An abnormal left ventricular ejection fraction (EF<55%)
6. History of a severe adverse reaction to beta blockers or calcium channel blockers (prior minor intolerance or ineffectiveness not exclusion)
7. Use of existing medication that has an unsafe drug--drug interaction with beta blockers or calcium channel blockers
8. Refusal to take beta blockers or calcium channel blockers
9. Resting systolic blood pressure <100 mmHg or heart rate <50 beats per minute
10. Inability to provide an informed consent, including an inability to speak, read, or understand English or Spanish
11. A hearing impairment that won't allow for a typical verbal conversation or a visual impairment that won't allow for reading of the written consent
12. A potentially vulnerable subject (including pregnant women, prisoners, economically and educationally disadvantaged, decisionally impaired, and institutionalized individuals)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2024-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Tremmel, MD, MS, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shaw LJ, Peterson ED, Shaw LK, Kesler KL, DeLong ER, Harrell FE Jr, Muhlbaier LH, Mark DB. Use of a prognostic treadmill score in identifying diagnostic coronary disease subgroups. Circulation. 1998 Oct 20;98(16):1622-30. doi: 10.1161/01.cir.98.16.1622. PMID 9778327

RESULTS

PARTICIPANT FLOW:
Groups:
- Beta Blocker (Nebivolol): Participants receive oral beta blocker (nebivolol 2.5 mg) once a day for 30 days.
- Calcium Channel Blocker (Diltiazem): Participants receive oral calcium channel blocker (Diltiazem-SR 120 mg) once a day for 30 days.
- Placebo: Participants receive placebo once a day for 30 days.
Period: Overall Study
Arm/Group | Beta Blocker (Nebivolol) | Calcium Channel Blocker (Diltiazem) | Placebo
Started | 2 | 1 | 2
Had at Least 1 Post-baseline Visit | 2 | 1 | 1
Completed | 2 | 1 | 1
Not Completed | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Beta Blocker (Nebivolol) | Calcium Channel Blocker (Diltiazem) | Placebo | Total
Number analyzed (Participants) | 2 | 1 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 2 | 5
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 3
  Male | 0 | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2 | 4
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 2 | 2
  White | 1 | 0 | 0 | 1
  Other | 1 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 1 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Angina Score Assessed by the Seattle Angina Questionnaire (SAQ)
Description: Effectiveness of beta blockers and calcium channel blockers for reducing angina in patients with a Myocardial Bridge (MB) compared to placebo determined after 30 days on the study drug by a change in angina, as assessed by the Seattle Angina Questionnaire (SAQ). The SAQ assesses 5 domains: physical limitation, angina stability angina frequency, treatment satisfaction, and quality of life. Each domain score is normalized to a range of 0 to 100, with higher scores corresponding to better outcomes.
Time Frame: baseline and 30 days
Population: Participants with data at the respective time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Beta Blocker (Nebivolol) | Calcium Channel Blocker (Diltiazem) | Placebo
Number analyzed (Participants) | 2 | 1 | 2
score on a scale
  Physical limitation - baseline | 44.4 (24.4) | 62.2 (NA) — Standard deviation not calculable for n of 1 | 53.4 (15.6)
  Physical limitation - 30 days: number analyzed (Participants) | 2 | 1 | 1
  Physical limitation - 30 days | 53.6 (24.5) | 68.0 (NA) — Standard deviation not calculable for n of 1 | 17.8 (NA) — Standard deviation not calculable for n of 1
  Angina stability - baseline | 40 (0) | 40 (NA) — Standard deviation not calculable for n of 1 | 80 (20)
  Angina stability - 30 days: number analyzed (Participants) | 2 | 1 | 1
  Angina stability - 30 days | 50 (30) | 60 (NA) — Standard deviation not calculable for n of 1 | 20 (0)
  Angina frequency - baseline | 70 (0) | 60 (NA) — Standard deviation not calculable for n of 1 | 75 (25)
  Angina frequency - 30 days: number analyzed (Participants) | 2 | 1 | 1
  Angina frequency - 30 days | 80 (10) | 80 (NA) — Standard deviation not calculable for n of 1 | 30 (NA) — Standard deviation not calculable for n of 1
  Treatment satisfaction - baseline | 67.7 (8.9) | 100 (NA) — Standard deviation not calculable for n of 1 | 76.5 (5.85)
  Treatment satisfaction - 30 days: number analyzed (Participants) | 2 | 1 | 1
  Treatment satisfaction - 30 days | 64.7 (11.8) | 94.1 (NA) — Standard deviation not calculable for n of 1 | 29.4 (NA) — Standard deviation not calculable for n of 1
  Quality of life - baseline | 41.6 (25) | 41.7 (NA) — Standard deviation not calculable for n of 1 | 37.5 (20.9)
  Quality of life - 30 days: number analyzed (Participants) | 2 | 1 | 1
  Quality of life - 30 days | 54.1 (20.9) | 58.3 (NA) — Standard deviation not calculable for n of 1 | 25 (NA) — Standard deviation not calculable for n of 1

2. Secondary Outcome: Duke Treadmill Score by Risk Category
Description: Changes in exercise capacity will be measured by difference in exercise time increment between the groups. The Duke treadmill score is calculated as exercise time × (5 × ST-segment deviation) - (4 × exercise angina), with 0 = no angina, 1 = non-limiting angina, and 2 = exercise-limiting angina. Possible scores range from -25 (highest risk) to +15 (lowest risk). Scores are reported by the number of participants in each risk category: low risk (≥+5), moderate risk (-10 to +4) and high risk (≤-11) (Shaw, et al, 1998).
Time Frame: baseline, 30 days
Population: Participants with data at the respective time point
Measure: Count of Participants; unit: Participants
Arm/Group | Beta Blocker (Nebivolol) | Calcium Channel Blocker (Diltiazem) | Placebo
Number analyzed (Participants) | 2 | 1 | 2
Participants
  Low risk - baseline | 0 | 0 | 0
  Moderate risk - baseline | 2 | 1 | 2
  High risk - baseline | 0 | 0 | 0
  Low risk - 30 days: number analyzed (Participants) | 1 | 1 | 1
  Low risk - 30 days | 0 | 1 | 0
  Moderate risk - 30 days: number analyzed (Participants) | 1 | 1 | 1
  Moderate risk - 30 days | 1 | 0 | 0
  High risk - 30 days: number analyzed (Participants) | 1 | 1 | 1
  High risk - 30 days | 0 | 0 | 1

3. Secondary Outcome: Duke Treadmill Score
Description: The Duke treadmill score is calculated as exercise time × (5 × ST-segment deviation) - (4 × exercise angina), with 0 = no angina, 1 = non-limiting angina, and 2 = exercise-limiting angina. Possible scores range from -25 (highest risk) to +15 (lowest risk).
Time Frame: baseline, 30 days
Population: Participants with data at the respective time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Beta Blocker (Nebivolol) | Calcium Channel Blocker (Diltiazem) | Placebo
Number analyzed (Participants) | 2 | 1 | 2
score on a scale
  Baseline | 2.3 (2.35) | 3.0 (NA) — Standard deviation not calculable for n of 1 | 1.5 (4.95)
  30 days: number analyzed (Participants) | 1 | 1 | 1
  30 days | 2 (NA) — Standard deviation not calculable for n of 1 | 10 (NA) — Standard deviation not calculable for n of 1 | -11 (NA) — Standard deviation not calculable for n of 1

4. Secondary Outcome: Number of Participants With Cardiac Events
Description: Major adverse cardiovascular events include death, heart attack, coronary stent or bypass surgery, and stroke.
Time Frame: 30 days, 6 months
Population: Participants with data at the respective time point
Measure: Count of Participants; unit: Participants
Arm/Group | Beta Blocker (Nebivolol) | Calcium Channel Blocker (Diltiazem) | Placebo
Number analyzed (Participants) | 2 | 1 | 1
Participants
  30 days | 0 | 0 | 0
  6 months | 0 | 0 | 0

5. Secondary Outcome: Drug Adherence.
Description: Percentage of drug taken by participants, measured by pill count at the end of 30 days.
Time Frame: 30 days
Population: Participants with data through 30 days
Measure: Mean (Standard Deviation); unit: percentage of drug taken
Arm/Group | Beta Blocker (Nebivolol) | Calcium Channel Blocker (Diltiazem) | Placebo
Number analyzed (Participants) | 2 | 1 | 1
percentage of drug taken | 99.5 (0.5) | 100 (NA) — Standard deviation not calculable for n of 1 | 100 (NA) — Standard deviation not calculable for n of 1

6. Secondary Outcome: Number of Participants With Side Effects
Description: Patient self-reported side effects recorded in a diary to be turned in at 30 days. In addition, patients are requested to contact us regarding any serious side effects during the study. Finally, patients are asked about any side effects they experienced during their 30-day follow-up to ensure that symptoms are captured.
Time Frame: 30 days
Population: Participants with data at 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Beta Blocker (Nebivolol) | Calcium Channel Blocker (Diltiazem) | Placebo
Number analyzed (Participants) | 2 | 1 | 1
Participants | 0 | 0 | 0

7. Secondary Outcome: Treatment Course
Description: Number of participants who stayed on the study drug at the initial dose, stayed on the study drug at a different dose, switched to an alternate therapy, and/or underwent further cardiac testing.
Time Frame: 6 months
Population: Participants with data at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Beta Blocker (Nebivolol) | Calcium Channel Blocker (Diltiazem) | Placebo
Number analyzed (Participants) | 2 | 1 | 1
Participants
  Stayed on study drug at the initial dose | 2 | 0 | 0
  Stayed on study drug at a different dose | 0 | 1 | 0
  Switched to alternate therapy | 0 | 0 | 1
  Underwent further cardiac testing | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Beta Blocker (Nebivolol) | Calcium Channel Blocker (Diltiazem) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/2

LIMITATIONS AND CAVEATS:
Early termination led to a small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/38/NCT04130438/Prot_SAP_000.pdf